CLINICAL TRIAL: NCT06771024
Title: Effectiveness of Community Physical Exercise Program in Chronic Disease (CPEP - Chronic Disease), a Clinical Randomized Controlled Trial
Brief Title: Community Physical Exercise Program in Chronic Disease
Acronym: CPEPCD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Associação para o Desenvolvimento do Centro Académico de Investigação e Formação Biomédica do Algarv (Network)
Collaborators: Loulé Municipal Council (Unknown); Albufeira Municipal Council (Unknown); Universidade do Algarve (Other)
Responsible Party: Principal Investigator, Marta Cristina Soares Botelho, Assistant Researcher, Associação para o Desenvolvimento do Centro Académico de Investigação e Formação Biomédica do Algarv
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPEP-Chronic Disease
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis Pain; Myocardial Infarction (MI); Hypertension; Dyslipidemia; Diabetes Mellitus; Overweight , Obesity; Stroke
Keywords: Physical Exercise Program; Healthy Ageing; Cardiovascular Risk; Osteoarthritis; Multimorbility; Chronic Diseases; Diabetes Mellitus; Cerebrovascular risk
MeSH Terms: conditions — Myocardial Infarction; Hypertension; Dyslipidemias; Diabetes Mellitus; Overweight; Obesity; Stroke; Osteoarthritis; Chronic Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants are assigned for two groups in parallel and a pre and post-test analysis is performed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Physical Exercise Program Group (Experimental): The participants receive a twelve weeks of a supervised physical exercise program, based on aerobic and strength training.
  Interventions: Behavioral: Physical Exercise
- Control Group (No Intervention): Participants do not receive any intervention.

INTERVENTIONS:
Behavioral: Physical Exercise — The intervention include a personalized physical exercise program based on aerobic and strength training, with prior warm-up and post cool-down exercises. International/national exercise prescription guidelines will be applied for each clinical condition (cardio/cerebrovascular disease/risk, diabetes mellitus and osteoarthritis). The main exercise component consists of concurrent training, combining resistance and aerobic exercises. The aims are to enhance muscle strength and endurance, improve self-confidence, increase the ability to perform activities of daily living, maintain independence, and reduce cardiac demands during daily activities (as indicated by a lower heart rate-pressure product). Training intensity is monitored using heart rate (HR) sensors. Blood pressure, HR, peripheral oxygen saturation (SpO₂), perceived exertion (Modified Borg Scale - MBS), and other relevant events are recorded in a daily log.
  Arms: Community Physical Exercise Program Group

SUMMARY:
This study focuses on promoting physical activity (PA) through the implementation of a Community Physical Exercise Program for Chronic Diseases (CPEP-CD), targeting individuals aged 50 years and older with at least two of the following conditions: cardiovascular and/or cerebrovascular disease or risk (CVD), overweight, diabetes mellitus (DM), and musculoskeletal diseases. The primary objective is to improve muscle and cardiorespiratory health and well-being, while also contributing to a more objective and evidence-based exercise prescription for these pathological conditions.

Population ageing is a global challenge associated with an increased prevalence of chronic diseases that compromise quality of life (QoL). A sedentary lifestyle is linked to declines in muscle function and cardiorespiratory fitness and is considered a major risk factor for morbidity and mortality. Consequently, physical exercise is widely recommended as a key non-pharmacological intervention across multiple chronic diseases.

According to World Health Organization (WHO) guidelines, regular PA is a protective factor in the prevention and management of non-communicable diseases, including cardiovascular and cerebrovascular diseases and DM. In addition, PA provides mental health benefits, supports healthy weight maintenance, and enhances overall well-being. In adults, regular PA is associated with reductions in all-cause mortality, cardiovascular mortality, and the incidence of hypertension.

Within this context, the aim of this project is to implement a community-based physical exercise program for individuals with chronic disease and multimorbidity, focusing on CVD and cerebrovascular disease or risk, DM, and OA. The program integrates existing exercise prescription guidelines while personalizing exercise progression according to both disease-specific and multimorbidity profiles. The primary outcomes include improvements in cardiorespiratory fitness, muscular strength, bone health, functional capacity, and QoL. Additionally, through individualized training monitoring, this study seeks to establish an exercise prescription tailored to the most prevalent combinations of chronic diseases, thereby providing more objective and practical guidance for family physicians, exercise professionals, and rehabilitation specialists, and supporting more personalized and targeted exercise-based strategies for chronic disease prevention and management.

DETAILED DESCRIPTION:
The implementation of exercise programs in individuals with chronic disease is essential for modifying cardiovascular and metabolic risk factors. However, it is equally important to examine not only the direct effects of exercise on health and well-being outcomes, but also to quantify the most appropriate training load, particularly in the presence of multimorbidity.

This is a non-pharmacological clinical study with two parallel intervention groups and a pre-post study design. Participants allocated to the Exercise Group (EG) will undertake a 12-week supervised physical exercise program, while those in the Control Group (CG) will receive no intervention during the study period.

Both groups will be assessed at two time points: (1) baseline assessment (T0) and (2) post-intervention assessment after 12 weeks (T12). The Community Physical Exercise Program (CPEP) will last 12 weeks, with two sessions per week, each lasting 60 minutes. International and national exercise prescription guidelines will be applied for each clinical condition, namely cardiovascular and/or cerebrovascular disease or risk, diabetes mellitus, and osteoarthritis. All variables will be assessed and monitored by qualified health and exercise professionals using reliable and validated instruments and equipment.

The training sessions will combine cardiorespiratory exercises aimed at improving aerobic capacity with strength training, particularly resistance exercises, using body weight and auxiliary equipment. Training intensity zones will be individualized and defined according to each participant's baseline cardiorespiratory fitness test results and subjective perception of effort.

The sample will include individuals aged 50 years or older with at least one of the aforementioned chronic conditions. Participation will be voluntary, and recruitment will be conducted through dissemination materials placed in senior universities, institutions and associations, municipalities, parish councils, sports facilities, health centers, and other relevant public spaces.

The sampling process will consist of an initial phase of non-random purposive sampling, followed by a second phase using snowball sampling if necessary. Sample size was calculated using G*Power software (version 3.1.9.7), assuming a two-tailed α level of 0.05, an effect size of 0.5, statistical power of 80%, and an anticipated dropout rate of 15%. A total sample of 147 participants will be required, with 74 participants allocated to each group.

Cardiovascular risk screening will be conducted based on the presence of one or more of the following risk factors: hypertension, dyslipidemia, or smoking, in accordance with SCORE2 or SCORE2-OP. For the other pathological conditions, definitions and criteria will be used in accordance with the recommendations of European or American scientific societies.

Following the intervention, the expected outcomes include improvements in cardiorespiratory fitness, muscular strength and muscle function, bone health, joint pain, physical function, quality of life, biochemical parameters related to glycemic and lipid profiles, and body composition. Additionally, the study aims to quantify the average training load and its progression over the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥50 years;
* At least 2 of the following: Prior cardiovascular disease (>12 months); High cardiovascular risk (SCORE2 or SCORE2 O.P.); Post-stroke (ischemic or hemorrhagic) with treated etiology; Type 2 Diabetes (> 6 months, ADA); Osteoarthristis (clinical signs/symptoms, NICE); Overweight/Obesity (BMI ≥ 27 kg/m2).
* Autonomous walking.
* Able to provide informed consent.
* Stable medications for ≥ 3 months (related to diagnoses of interest).
* Physical activity below WHO recommendations.
* No contraindications to exercise (cardiovascular, cerebrovascular, respiratory, musculoskeletal) according to ACSS.

Exclusion Criteria:

* Moderate to severe cognitive impairment - Montreal Cognitive Assessment (MoCA).
* Type 2 Myocardial Infarction.
* Class III or IV angina (Canadian Cardiovascular Society).
* Class III or IV angina (New York Heart Association).
* Uncontrolled CVD: symptomatic arrhythmias with hemodynamic compromise; severe symptomatic aortic valve stenosis; uncontrolled symptomatic heart failure; endocarditis, pericarditis, or active myocarditis; acute aortic syndrome; suspected or known dissecting aneurysm; acute systemic infections.
* Pacemaker user.
* Neurological disorders affecting gait.
* Severe diabetes-related complications contraindicating exercise (poor metabolic control, diabetic foot, diabetic retinopathy, diabetic nephropathy, and diabetic autonomic neuropathy).
* Recent use of insulin or sulphonylureas (< 3 months).
* Untreated stroke etiology: indication for revascularization; non-anticoagulated atrial fibrillation; intracranial atherosclerotic occlusive disease.
* Musculoskeletal or ocular conditions preventing strength training (acute herniated disc, fractures, recent spinal surgery, glaucoma with elevated intraocular pressure).
* Terminal illness.
* Inability to understand basic oral or written Portuguese.
* Participation in supervised dietary intervention.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Peak Oxygen Uptake (VO2peak) | 12 weeks
  Significant increase in Peak Oxygen Uptake (VO2peak). Higher VO2peak means better cardiorespiratory function. The VO2peak will be evaluated through the exercise cardiorespiratory test with progressive increase of the external load in a cycle ergometer.
Change in First Ventilatory Threshold (VT1 - VO2) | 12 weeks
  Significant increase in First Ventilatory Threshold (VT1 - VO2). Higher VT1 means better cardiorespiratory function. The VT1 will be evaluated through the exercise cardiorespiratory test with progressive increase of the external load in a cycle ergometer.
Change in Respiratory Compensation Point (RCP - VO2) | 12 weeks
  Significant increase in Respiratory Compensation Point (RCP - VO2). Higher RCP means better cardiorespiratory function. The RCP will be evaluated through the exercise cardiorespiratory test with progressive increase of the external load in a cycle ergometer.
Change in peak torque of quadriceps and hamstring muscles | 12 weeks
  A significant increase in peak torque (N/m). Peak torque of the quadriceps and hamstring muscles will be measured using a fixed dynamometer with concentric-concentric actions at an angular velocity of 60° per second, during five maximal repetitions of knee extension and flexion for each knee.
Change in work of quadriceps and hamstring muscles | 12 weeks
  A significant increase in work per repetition (N/m). Work of the quadriceps and hamstring muscles will be measured using a fixed dynamometer with concentric-concentric actions at an angular velocity of 60° per second, during five maximal repetitions of knee extension and flexion for each knee.
Change in power of quadriceps and hamstring muscles | 12 weeks
  A significant increase in power per repetition (W). Peak torque of the quadriceps and hamstring muscles will be measured using a fixed dynamometer with concentric-concentric actions at an angular velocity of 60° per second, during five maximal repetitions of knee extension and flexion for each knee.

SECONDARY OUTCOMES:
Change in lower limb functionality (number of repetions) | 12 weeks
  A significant increase in lower limb functional performance, reflected by an increased number of repetitions, is expected. Lower limb functionality will be assessed using the 30-Second Sit-to-Stand Test (30STS).
Change in functional mobility (seconds) | 12 weeks
  A significant improvement in functional mobility, reflected by a decrease in the time required to complete the Timed Up and Go (TUG) test, is expected. The TUG test will be performed with participants rising from a standard chair, walking 3 meters at a comfortable pace, turning, returning to the chair, and sitting down.
Change in Oscillation of the Center of Pressure | 12 weeks
  The balance analysis will be carried out using an AMTI® force platform, which will allow determining the displacement and oscillation of the static center of pressure (CP) with participants in 2 conditions: eyes open and eyes closed (duration of 30 seconds for each assessment).
Change in Health-Related Quality of Life | 12 weeks
  A significant improvement in health-related quality of life (HRQoL) is expected. HRQoL will be assessed using the EQ-5D-5L questionnaire (EuroQol Group), which evaluates five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension comprises five levels of severity, ranging from 1 (no problems) to 5 (extreme problems or inability). The EuroQol Visual Analogue Scale (EQ VAS) will also be used.
Change in Hand Grip Strength | 12 weeks
  Significant increase in hand grip strength (kg). Higher hand grip strength is correlated with higher functional status. Maximum handgrip strength will be measured with the Lafayette Digital and Dynamometer 5030D1 manual digital dynamometer on the dominant upper limb.
Change in Weight | 12 weeks
  Significant decrease in weight (kg). Higher values of weight mean poor body composition and health. The weight will be measured using the bioimpedance technique.
Change in body mass index | 12 weeks
  Significant decrease in body mass index (kg/m2). Higher values of body mass index mean poor body composition and health. The body mass index will be measured using the bioimpedance technique.
Change in fat mass | 12 weeks
  Significant decrease in fat mass (kg and %)). Higher values of fat mass mean poor body composition and health. The fat mass will be measured using the bioimpedance technique.
Change in fat-free mass | 12 weeks
  Significant increase in fat-free mass (kg and %). Higher values of fat-free mass mean better body composition and health. The fat-free mass will be measured using the bioimpedance technique.
Change in fat mass index | 12 weeks
  Significant decrease in fat mass index (kg/m2). Higher values of fat mass index mean poor body composition and health. The fat mass index will be measured using the bioimpedance technique.
Change in fat-free mass index | 12 weeks
  Significant increase in fat-free mass index (kg/m2). Higher values of fat-free mass index mean better body composition and health. The fat-free mass index will be measured using the bioimpedance technique.
Change in muscle mass index | 12 weeks
  Significant increase in muscle mass index (kg/m2). Higher values of muscle mass index mean better body composition and health. The muscle mass index will be measured using the bioimpedance technique.
Monitoring phase angle | 12 weeks
  Keep the phase angle within normal limits for the age. The phase angle will be measured using the bioimpedance technique.
Change in fat visceral fat | 12 weeks
  Significant decrease in visceral fat (L). Higher values of visceral fat mean poor body composition and health. The visceral fat will be measured using the bioimpedance technique.
Change in abdominal circumference | 12 weeks
  Significant decrease in abdominal circumference (cm). Higher values of abdominal circumference mean poor body composition and health. The abdominal circumference will be measured using measure tape, according to the STEPS Manual of the World Health Organization.
Changes in Total cholesterol (mg/dL) - Lipid Profile | 12 weeks
  Total cholesterol (mg/dL) will be measured taking a sample blood which will be analysed by the COBAS b 101 system.
Changes in Triglycerides (mg/dL) - Lipid Profile | 12 weeks
  Triglycerides (mg/dL) will be measured taking a sample blood which will be analysed by the COBAS b 101 system.
Changes in High-density lipoprotein (HDL) cholesterol (mg/dL) - Lipid Profile | 12 weeks
  High-density lipoprotein (HDL) cholesterol (mg/dL) will be measured taking a sample blood which will be analysed by the COBAS b 101 system.
Changes in Low-density lipoprotein (HDL) cholesterol (mg/dL) - Lipid Profile | 12 weeks
  Low-density lipoprotein (HDL) cholesterol (mg/dL) will be measured taking a sample blood which will be analysed by the COBAS b 101 system.
Changes in Glicemic Profile (HbA1c) | 12 weeks
  Glicemic Profile will be measured by COBAS b 101 system, taking a sample blood which will be analysed for Glycated Hemoglobin (HbA1c).
Change in contraction time of bíceps femoris, tibial anterior and lateral gastrocnemius bi-lateral | 12 weeks
  Significant decrease in contraction time (ms) of bíceps femoris, tibial anterior and lateral gastrocnemius. Higher contraction time means poor muscle function. The contraction time will be measured by a tensiomyography system TMG S2. Tensiomyography assesses contractile properties of an isolated muscle by measuring a few parameters in response to a twitch contraction.
Change in radial muscle belly displacement of bíceps femoris, tibial anterior and lateral gastrocnemius bi-lateral | 12 weeks
  Significant decrease in radial muscle belly displacement (mm) of bíceps femoris, tibial anterior and lateral gastrocnemius. Higher radial muscle belly displacement means poor muscle function and muscle atrophy. The radial muscle belly displacement will be measured by a tensiomyography system TMG S2. Tensiomyography assesses contractile properties of an isolated muscle by measuring a few parameters in response to a twitch contraction.
Change in latence time of bíceps femoris, tibial anterior and lateral gastrocnemius bi-lateral | 12 weeks
  Significant decrease in latence time (ms) of bíceps femoris, tibial anterior and lateral gastrocnemius. Higher latence time means poor muscle function. The latence time will be measured by a tensiomyography system TMG S2.
  Tensiomyography assesses contractile properties of an isolated muscle by measuring a few parameters in response to a twitch contraction.
Change in bone mineral density (BMD) | 12 weeks
  Significant increase in bone mineral density (BMD) (g/cm2) and improvement in T-score and Z-score. A higher BMD indicates reduced bone fragility. BMD will be assessed using a Radiofrequency Echographic Multi-Spectrometry (REMS) device at the lumbar spine and femoral neck.
Change in Osteoarthritis (OA) Symptoms and Function | 12 weeks
  A significant reduction in osteoarthritis (OA) symptoms and an improvement in physical function are expected. Symptoms and disability in knee and hip OA will be assessed using the Western Ontario and McMaster Universities Arthritis Index (WOMAC), which comprises pain, stiffness, and physical function subscales. Each item is scored on a scale from 0 to 4, with lower scores indicating fewer symptoms and better functional status.

OTHER OUTCOMES:
Monitoring Diabetic Peripheral Neuropathy -DPN | 0
  To assess the presence and level of severity of DPN, the Michigan Neuropathy Screening Instrument (MNSI) will be used. The MNSI is divided into two parts: questionnaire (Q) and physical examination (FE). The following cutoffs are used at Q-MNSI ≥ 4.0 and/or at EF-MNSI ≥ 2.5.

CONTACTS AND LOCATIONS:
Locations (1):
- Algarve Biomedical Center, Faro, Algarve, Portugal

IPD SHARING:
Plan to Share IPD: Undecided